CLINICAL TRIAL: NCT04580121
Title: An Open-Label, Multi-Center, Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RO7283420 as a Single Agent in Hematologic and Molecular Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: A Dose Escalation and Expansion Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RO7283420.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: WP42004; 2020-000216-30 (EudraCT Number)
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — tocilizumab; Dasatinib; Dexamethasone; Acetaminophen; Diphenhydramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: Single Participant Dose Escalation (Experimental): Participants from Group I will receive escalating doses of RO7283420, once every 3 weeks (Q3W) starting on Cycle 1, Day 1 (C1D1) for up to 6 cycles with a starting dose of 0.15mg.
  Interventions: Drug: RO7283420; Drug: Tocilizumab; Drug: Dasatinib; Drug: Dexamethasone; Drug: Paracetamol/acetaminophen; Drug: Diphenhydramine
- Part B: Multiple Participant Dose Escalation (Experimental): Multiple-participant cohorts of >= 3 participants will be enrolled for dose escalation for Group I and Group II independently. Participants will be administered a starting dose of 0.15 mg or highest dose administered in Part A. Each participant will receive up to 6, 9, and 18 cycles of treatment with RO7283420, when treated with Q3W, every-2-weeks (Q2W), or once-a-week (QW) dosing regimens, respectively to determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D). Additionally, step-up dosing regimens with more frequent administrations of RO7283420 during cycle 1 will be evaluated.
  Interventions: Drug: RO7283420; Drug: Tocilizumab; Drug: Dasatinib; Drug: Dexamethasone; Drug: Paracetamol/acetaminophen; Drug: Diphenhydramine
- Part C: Dose Expansion (Experimental): Participants will receive the respective RP2D for Group I and Group II.
  Interventions: Drug: RO7283420; Drug: Tocilizumab; Drug: Dasatinib; Drug: Dexamethasone; Drug: Paracetamol/acetaminophen; Drug: Diphenhydramine

INTERVENTIONS:
Drug: RO7283420 — RO7283420 will be administered to participants by intravenous (IV) infusion Q3W at a starting dose of 0.15mg. Starting dose levels (double step-up regimen, Q3W) for SC injections was the same as the highest dose levels that have been cleared in the IV double step-up cohorts at that timepoint. Each participant will receive up to 6, 9, and 18 cycles of treatment with RO7283420, when treated with Q3W, Q2W, or QW dosing regimens, respectively.
  Arms: Part A: Single Participant Dose Escalation; Part B: Multiple Participant Dose Escalation
Drug: RO7283420 — RO7283420 at RP2D will be administered by IV infusion or SC injection as per dosing schedule determined in Part B.
  Arms: Part C: Dose Expansion
Drug: Tocilizumab — Tocilizumab will be administered as an IV infusion 8 mg/kg (for participants with a weight of 30 kg and above) and 12 mg/kg (for participants with a weight of less than 30 kg). Tocilizumab will be given as rescue medication.
  Other Names: Actemra, RoActemra
Drug: Dasatinib — Dasatinib 100 mg film-coated tablets will be administered daily until symptom resolution (up to 100 mg twice daily [BID] for a maximum 3 days); orally. Dasatinib will be given as rescue medication.
Drug: Dexamethasone — 20 mg IV of dexamethasone will be administered as pre-medication at least 60 minutes prior to the all RO7283420 infusions or injections during cycle 1.
Drug: Paracetamol/acetaminophen — 500 or 1000 mg of paracetamol/acetaminophen will be administered orally or by IV as pre-medication at least 30 minutes prior to each RO7283420 infusion or injection.
Drug: Diphenhydramine — 25 mg or 50 mg of diphenhydramine will be administered orally or by IV as pre-medication at least 30 minutes prior to each RO7283420 infusion or injection.

SUMMARY:
This open-label, entry-into-human (EIH) study will evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics of RO7283420. Escalating doses of RO7283420 will be administered to participants with Acute Myeloid Leukemia (AML) in order to determine the maximum tolerated dose (MTD) and/or recommended Phase II dose (RP2D).

DETAILED DESCRIPTION:
The study will include AML participants with measurable disease, for whom standard-of-care (SOC) is not available. Two Groups of AML participants will be included in this study:

* Group I participants will have hematologic relapse/refractory disease defined as participants not in complete remission (CR) or complete remission with incomplete hematologic recovery (CRi).
* Group II participants will have molecular relapse/persistent disease (participants with a CR or CRi, and a positive MRD based on local multi-parameter flow cytometry (MFC) or molecular assessment).

The study consists of three parts:

* Part A (single-participant dose escalation cohorts) - single participants from Group I will receive increment-based escalating doses until a Grade >=2 AE related to RO7283420 or a clear pharmacodynamic effect
* Part B (multiple-participant dose escalation cohorts) - multiple-participant cohorts of >=3 participants will be enrolled for dose escalation for Group I and Group II independently.
* Part C (dose expansion) - participants will receive the respective identified RP2D for that group.

The treatment period for each participant will be up to 7 months with a maximum number of cycles depending on the dosing frequency the participant receives. Each participant will receive up to 6, 9, and 18 cycles of treatment with RO7283420, when treated with Q3W, every-2-weeks (Q2W), or once-a-week (QW) dosing regimens, respectively. Additional 3, 5, or 9 cycles may be administered for the Q3W, Q2W, and QW dosing regimens, respectively, in case the participants have achieved at least partial remission (PR).

ELIGIBILITY:
Inclusion Criteria:

* With confirmed diagnosis of primary or secondary AML according to WHO classification 2016, with measurable disease. Eligible participants need to have received standard-of-care (SOC) and have no other SOC options available Participants who are not willing to receive SOC will be not eligible. Two groups of participants (Group I - hematologic relapsed/refractory and Group II - molecular relapsed/refractory) will be included
* Participants who have received hematopoietic stem cell transplant (HSCT) must have the HSCT performed ≥ 90 days prior to the first dose of RO7283420 on Cycle 1 Day 1, having demonstrated hematological engraftment and do not have an active Graft versus Host Disease, not requiring immunosuppressive treatment (including but not limited to cyclosporine, tacrolimus, sirolimus, and mycophenolate), which must be stopped at least 28 days prior to the first dose of RO7283420 on Cycle 1 Day 1
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Peripheral blast counts =< 20,000/mm3 on Cycle 1 Day 1 prior to the first dosing
* Confirmed genotype of HLA-A*02
* Adequate renal (a creatinine clearance of >=50 mL/min as calculated according to the Cockroft-Gault formula) and adequate liver test results
* Male or female participants agree to use contraception and the abstinence requirements to prevent exposure of an embryo to the study treatment

Exclusion Criteria:

* Acute promyelocytic leukemia (APL)
* Core Binding Factor (CBF)-AML Note: participants with r/r CBF-AML after at least 2 salvage attempts can be enrolled into the study
* Group II only: participants with normal karyotype and a favorable molecular profile according to ELN guideline 2017
* Participants with active bacterial, fungal or viral infection considered by the Investigator to be clinically uncontrolled or of unacceptable risk upon the induction of neutropenia (i.e. participants who are or should be on antimicrobial agents for the treatment of active infection)
* Grade >= 2 glomerular proteinuria at screening or on Cycle 1 Day 1 prior to the first dosing.
* Another primary malignancy (other than AML) that requires active therapy. Adjuvant hormonal therapy is allowed
* Clinical evidence or history of central nervous system (CNS) leukemia
* Presence of extramedullary disease at screening
* Current or past history of CNS disease, such as stroke, CNS inflammation, epilepsy, CNS vasculitis, or neurodegenerative disease
* Participants who have a history of clinically significant liver disease, including liver cirrhosis (e.g. Child-Pugh class B and C) or participants who have a history of active or chronic infectious hepatitis unless serology demonstrates clearance of infection
* Participants who might refuse to receive blood products and/or have known hypersensitivity to any of the components of RO7283420, tocilizumab, or dasatinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2023-08-09 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | From baseline up to 9 months
Percentage of Participants with Dose-Limiting Toxicities (DLTs) | From baseline up to 28 days
Recommended Phase II Dose (RP2D) | From baseline up to 7 months

SECONDARY OUTCOMES:
Maximum Reduction (%) from Baseline in Blast Count in Peripheral Blood and/or Bone Marrow (Group I Dose Escalation Cohorts only) | From baseline up to 7 months
Percentage of Participants who Achieve a Response | From baseline up to approximately 4 years
  Defined by ELN 2017 recommendations, i.e., complete remission (CR), complete remission with incomplete hematologic recovery (CRi), complete remission with absence of measurable residual disease (CRMRD-), and partial remission (PR).
Transfusion Independence | From baseline up to 7 months
Event-free Survival (EFS) | From baseline to the time to progression, relapse, death from any cause, or start of a new treatment (up to approximately 4 years)
Duration of Response (DoR) | From first occurrence of a documented response until the time of documented relapse, disease progression or death from any cause, whichever occurs first (up to approximately 4 years)
Time to Hematological Relapse (Group II Only) | From baseline until the time of documented hematological relapse
Early Mortality Rate | From baseline to Day 30, and to Day 60
Progression-free Survival (PFS) | From Cycle 1 Day 1 to the first occurrence of documented disease progression, or death from any cause, whichever occurs first (up to approximately 4 years)
Number of MRD (Measurable Residual Disease) Negative Participants over time According to Local MRD Assessment | From baseline up to 7 months
Area Under the Curve (AUC) of RO7283420 | Day 1, 2, 3, 8, 15 of Cycle 1 (each cycle is 21 days); Day 1, 2, 3, 8 of Cycle 2 only in case of triple step-up dosing; Day 1 of Cycle 2-9 (Q3W), 2-14 (Q2W), 2-27 (QW); end of treatment visit.
Maximum Concentration (Cmax) of RO7283420 | Day 1, 2, 3, 8, 15 of Cycle 1 (each cycle is 21 days); Day 1, 2, 3, 8 of Cycle 2 only in case of triple step-up dosing; Day 1 of Cycle 2-9 (Q3W), 2-14 (Q2W), 2-27 (QW); end of treatment visit.
Minimum Concentration (Cmin) of RO7283420 | Day 1, 2, 3, 8, 15 of Cycle 1 (each cycle is 21 days); Day 1, 2, 3, 8 of Cycle 2 only in case of triple step-up dosing; Day 1 of Cycle 2-9 (Q3W), 2-14 (Q2W), 2-27 (QW); end of treatment visit.
Clearance (Cl) of RO7283420 | Day 1, 2, 3, 8, 15 of Cycle 1 (each cycle is 21 days); Day 1, 2, 3, 8 of Cycle 2 only in case of triple step-up dosing; Day 1 of Cycle 2-9 (Q3W), 2-14 (Q2W), 2-27 (QW); end of treatment visit.
Volume (V) of RO7283420 | Day 1, 2, 3, 8, 15 of Cycle 1 (each cycle is 21 days); Day 1, 2, 3, 8 of Cycle 2 only in case of triple step-up dosing; Day 1 of Cycle 2-9 (Q3W), 2-14 (Q2W), 2-27 (QW); end of treatment visit.
Half-life (T1/2) of RO7283420 | Day 1, 2, 3, 8, 15 of Cycle 1 (each cycle is 21 days); Day 1, 2, 3, 8 of Cycle 2 only in case of triple step-up dosing; Day 1 of Cycle 2-9 (Q3W), 2-14 (Q2W), 2-27 (QW); end of treatment visit.
Incidence and Titer of Anti-drug Antibodies (ADA) against RO7283420 | Day 1, 8, 15 of Cycle 1 (each cycle is 21 days); Day 1 and 8 of Cycle 2, Day 1 of Cycle 3-9 (Q3W), 3-14 (Q2W), 3-27 (QW); at end of treatment visit

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (23):
- United States (2):
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (2):
  - Peter MacCallum Cancer Centre; Medical Oncology, Melbourne, Victoria
  - The Alfred, Melbourne, Victoria
- Princess Margaret Cancer Center, Toronto, Ontario, Canada
- Rigshospitalet; Hæmatologisk Klinik, Klinisk Afprøvnings Team KAT, København Ø, Denmark
- France (2):
  - Institut Paoli Calmettes; Departement D' Onco-Hematologie, Marseille
  - Hopital De Haut Leveque; Hematologie Clinique, Pessac
- Germany (2):
  - Uniklinikum "Carl Gustav Carus"; Med. Klinik 1; Hämatologie, Zelltherapie und Medizinische Onkologie, Dresden
  - Klinikum der Universität München, Campus Großhadern; Medizinische Klinik und Poliklinik III, München
- Italy (3):
  - ASST PAPA GIOVANNI XXIII; Ematologia, Bergamo, Lombardy
  - Istituto Clinico Humanitas;U.O. Oncologia Medica Ed Ematologia, Rozzano, Lombardy
  - Ospedale Santa Chiara; Unita Operativa Di Ematologia, Pisa, Tuscany
- Spain (5):
  - Institut Catala d?Oncologia Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitari Vall d'Hebron; Servicio de Hematologia, Barcelona
  - Hospital Clínic i Provincial; Servicio de Hematología y Oncología, Barcelona
  - Hospital Univ. 12 de Octubre; Servicio de Hematologia, Madrid
  - Hospital Universitario la Fe; Servicio de Hematologia, Valencia
- Taiwan (3):
  - China Medical University Hospital; Oncology and Hematology, Taichung
  - National Cheng Kung University Hospital; Oncology, Tainan
  - National Taiwan Universtiy Hospital; Division of Hematology, Taipei
- United Kingdom (2):
  - Churchill Hospital, Oxford
  - Royal Marsden NHS Foundation Trust, Sutton

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Hutchings M, Korfi K, Montesinos P, Santoro A, Hou HA, Martinez-Sanchez P, Vives S, Galimberti S, Chen TY, Frigeni M, Garciaz S, Salamero Garcia O, Yeh SP, Yee K, Esteve J, Bajel A, Fleming S, Bretz AC, Attig J, Sun M, Nassiri S, Rutishauser T, Klein C, Ma YM, Schnetzler G, Vauleon S, Yu H, Barata T, Richard M, Simon S, Hinton H, Keshelava N, Subklewe M. Dose escalation study of the HLA-A2-WT1 CD3 bispecific antibody RO7283420 in relapsed/refractory acute myeloid leukemia. Blood Neoplasia. 2025 May 11;2(3):100110. doi: 10.1016/j.bneo.2025.100110. eCollection 2025 Aug. PMID 40746940
- [Derived] Augsberger C, Hanel G, Xu W, Pulko V, Hanisch LJ, Augustin A, Challier J, Hunt K, Vick B, Rovatti PE, Krupka C, Rothe M, Schonle A, Sam J, Lezan E, Ducret A, Ortiz-Franyuti D, Walz AC, Benz J, Bujotzek A, Lichtenegger FS, Gassner C, Carpy A, Lyamichev V, Patel J, Konstandin N, Tunger A, Schmitz M, von Bergwelt-Baildon M, Spiekermann K, Vago L, Jeremias I, Marrer-Berger E, Umana P, Klein C, Subklewe M. Targeting intracellular WT1 in AML with a novel RMF-peptide-MHC-specific T-cell bispecific antibody. Blood. 2021 Dec 23;138(25):2655-2669. doi: 10.1182/blood.2020010477. PMID 34280257